CLINICAL TRIAL: NCT05677048
Title: Feasibility Study: IGNITE-TX (Identifying Individuals for Genetic Testing & Treatment) Intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-0712; FP00015533 (Other Grant/Funding Number: Foundation for Women's Cancer); NCI-2022-10573 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-12-14; First posted 2023-01-10 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Gynecologic Cancer; Ovary Cancer; Pancreatic Cancer; Breast Cancer; Lynch Syndrome; Hereditary Breast and Ovarian Cancer Syndrome; Colon Cancer; Endometrial Cancer; Uterus Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Pancreatic Neoplasms; Breast Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis; Hereditary Breast and Ovarian Cancer Syndrome; Colonic Neoplasms; Endometrial Neoplasms; Uterine Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Standard of Care Group) (No Intervention): Participants (probands, those with a hereditary cancer syndrome) are sent a family letter to share with relatives. The letter contains information about hereditary cancer syndromes and encourages relatives to participate in the study and to get genetic testing.
  Relatives of probands randomized to the usual care arm will have access to the family letter if probands decide to share it with them, and will receive study surveys. The letter contains information about hereditary cancer syndromes and encourages relatives to participate in the study and to get genetic testing
- Group 2 (Free genetic testing and counseling group) (Experimental): Enrolled relatives will receive a letter and baseline survey with information to contact the tele-genetics company to arrange free genetic counseling and testing. This letter will be given to the relatives directly by the study
  Interventions: Behavioral: Free genetic testing and counseling group; Behavioral: IGNITE-TX Group; Behavioral: IGNITE-TX and free genetic testing and counseling group
- Group 3 (IGNITE-TX Group) (Experimental): Relatives of probands randomized to the IGNITE-TX intervention will receive a family letter after enrollment and baseline survey with their personal access codes (not to be shared) to the IGNITE-TX "Hub" (access online educational material through a platform). Relatives will have also access services of a family genetic navigator. Study investigators and navigators will not directly provide genetic counseling and/or testing in this arm
  Interventions: Behavioral: Free genetic testing and counseling group; Behavioral: IGNITE-TX Group; Behavioral: IGNITE-TX and free genetic testing and counseling group
- Group 4 (IGNITE-TX and free genetic testing and counseling group) (Experimental): Relatives randomized to this arm will receive a family letter after enrollment and baseline survey with their personal access codes (not to be shared) to the IGNITE-TX "Hub" (access online educational material through a platform) and information to contact the tele genetics company. This arm will receive both the IGNITE-TX Intervention and access to free genetic testing and counseling services, as well as access to assistance from family genetic navigator
  Interventions: Behavioral: Free genetic testing and counseling group; Behavioral: IGNITE-TX Group; Behavioral: IGNITE-TX and free genetic testing and counseling group

INTERVENTIONS:
Behavioral: Free genetic testing and counseling group — Option to access no-cost telegenetic counseling and genetic testing
  Arms: Group 2 (Free genetic testing and counseling group); Group 3 (IGNITE-TX Group); Group 4 (IGNITE-TX and free genetic testing and counseling group)
Behavioral: IGNITE-TX Group — Access online educational materials through the IGNITE-TX platform and receive assistance from a family genetic navigator
  Arms: Group 2 (Free genetic testing and counseling group); Group 3 (IGNITE-TX Group); Group 4 (IGNITE-TX and free genetic testing and counseling group)
Behavioral: IGNITE-TX and free genetic testing and counseling group — Option to access no-cost telegenetic counseling and genetic testing, access to online educational materials through the IGNITE-TX platform, and assistance from a family genetic navigator
  Arms: Group 2 (Free genetic testing and counseling group); Group 3 (IGNITE-TX Group); Group 4 (IGNITE-TX and free genetic testing and counseling group)

SUMMARY:
This is a community-based study requiring participant-self-enrollment, that can help to increase the rates of genetic testing among the family members of people who have been diagnosed with a hereditary cancer syndrome. The two main factors in this study are the IGNITE-TX intervention (website and navigator) and the free genetic counseling and testing.

The IGNITE-TX Intervention is an innovative multi-modal intervention, with two components: a) interactive web "IGNITE-TX Hub" and b) genetic family navigators.

DETAILED DESCRIPTION:
Primary Objectives:

The primary objectives of this study are to assess the study feasibility by estimating:

1. The enrollment of probands and (ARRs) at-risk relatives over a 6-month period
2. The response rate to baseline and follow-up surveys by probands
3. The response rate to baseline and follow-up surveys by (ARRs) at-risk relatives

Secondary Objectives:

The secondary objectives of this study are to:

1. Measure (ARR) at-risk relatives completion of (CGT) cascade genetic testing among different study arms.
2. Measure the proportion of enrolled (ARRs) at-risk relatives who make an informed decision about (CGT) cascade genetic testing.
3. Measure the (ARR) at-risk relatives readiness for (CGT) cascade genetic testing
4. Measure proband and (ARR) at-risk relatives change in genetics knowledge
5. Measure proband readiness to communicate results of genetic testing with (ARR) at-risk relatives Secondary objectives in this feasibility study will be primary objectives in a larger study. This feasibility study is not powered to assess these objectives. Including them in this feasibility study will allow for assessment of our measurement tools (surveys from primary objectives) and offer insight into how the intervention may impact cascade genetic testing when implemented on a larger scale

Exploratory Objectives:

The exploratory objectives in this study are to estimate:

1. The average website traffic of the IGNITE-TX "Hub" and module completion
2. The average utilization of family genetic navigators by participants
3. Estimate the intra-familial correlation (IFC) for (ARR) at-risk relatives completion of (CGT) cascade genetic testing
4. Assess satisfaction with IGNITE-TX website modules and genetic navigator The exploratory objectives will allow for further evaluation of the IGNITE-TX website modules and navigator and understand how families with multiple (ARR)at-risk relatives respond to the intervention.

ELIGIBILITY:
Probands

Inclusion Criteria:

1. 18 years of age or older
2. Speaks and/or reads English or Spanish
3. Has known deleterious/pathogenic mutation or suspected deleterious/pathogenic variant in BRCA1 or BRCA2 (HBOC) or MLH1, MSH2, MSH6, PMS2, or EPCAM (LS)
4. Has access to the internet or phone and can send and receive email and/or text messages at a US telephone number
5. Has at least one at-risk relative who meets inclusion criteria for first-degree relative

Exclusion Criteria:

1. Has no at-risk relatives meeting inclusion criteria
2. Has negative germline genetic testing or only variant of uncertain significance
3. Unwilling or unable to provide consent 4.2. AT-RISK RELATIVES (ARR)

Inclusion Criteria:

1. 18 years of age or older
2. Speaks and reads English or Spanish
3. Resides in the United States
4. Can provide proof of deleterious/suspected deleterious HBOC or LS variant present in a first degree relative (biological mother or father, biological child, or full sibling)
5. Has access to internet or phone and can send and receive email and/or text messages at a US telephone number

Exclusion Criteria:

1. Unwilling or unable to provide consent
2. Reports no known HBOC or LS variant within the family
3. Has already been tested for the variant identified in the proband
4. Already listed as an ARR for another proband

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2023-04-14 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Measure enrollment of probands and at-risk relatives over a 6-month period | Up to 6 months
Measure response rate to baseline and follow-up surveys by probands and at-risk relatives | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jose Rauh-Hain, MD,MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org